CLINICAL TRIAL: NCT02381951
Title: Spinal Cord Stimulation in the Treatment of Parkinson's Disease
Acronym: STIMUPARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-A01356-41
Record Dates: First submitted 2015-03-03; First posted 2015-03-06 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2017-07

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spinal cord stimulation (Experimental)
  Interventions: Device: spinal cord stimulation (St Jude Medical)

INTERVENTIONS:
Device: spinal cord stimulation (St Jude Medical) — implantation of a spinal cord neurostimulation system : St Jude Medical Octrode 3183 (R) peridural lead connected to a St Jude Medical EonC (R) primary cell IPG

SUMMARY:
Parkinson's disease affects between 100'000 and 150'000 people in France. Drug therapy (L-Dopa and other drugs) is effective to improve motor symptoms but after an initial 'honeymoon period' lasting a few years, motor symptoms reoccur in most patients, impairing gait and walking.

Spinal cord stimulation is currently an important therapeutic option in the treatment of neuropathic pain. Experimental and limited clinical data suggest that this technique might also be used to alleviate motor symptoms and improve walking in Parkinsons patients.

This exploratory study aims at measuring the benefits of spinal cord stimulation on the walking capacity of a small number of Parkinsons patients who are not adequately improved by drug therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease since more than 5 years
* Walking disorder with freezing episodes, insufficiently alleviated by oral dopaminergic therapy and/or physiotherapy

Exclusion Criteria:

* Atypical Parkinson-like syndrome (e.g. progressive supranuclear palsy)
* Cognitive impairment (MMSE<24)
* Psychiatric disease
* Contraindication of surgery
* Neuropathic pain in the lower limb or lumbar region

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2017-04-25 (Actual)

PRIMARY OUTCOMES:
improvement in walking capacity | 2 months
  "stand-walk-sit" test : time to complete the test : difference between scores pre-implantation and 2 month post-implantation of stimulator

SECONDARY OUTCOMES:
freezing episodes : reduction of frequency | 2 months
  "stand-walk-sit" test : total number of freezing episodes during the test : difference between scores pre-implantation and 2 month post-implantation of stimulator
freezing episodes : reduction of cumulated time | 2 months
  "stand-walk-sit" test : cumulated time of freezing episodes during the test : difference between scores pre-implantation and 2 month post-implantation of stimulator
improvement in motor score of MultiDimentionalScaling-UPDRS scale | 2 months
  percentage of improvement in the motor score (part III of scale) of MultiDimentionalScaling-UPDRS scale, between score pre-implantation and score 2 months post-implantation of stimulator
improvement in "freezing of gait" score | 2 months
  percentage of improvement in the "freezing of gate" score, between score pre-implantation and score 2 months post-implantation of stimulator
improvement in quality of life score | 2 months
  improvement in PDQ 39 quality of life score between pre-implantation visit and 2 months post-implantation of stimulator

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique A. de Rothschild, Paris, France

REFERENCES:
- [Result] Hubsch C, D'Hardemare V, Ben Maacha M, Ziegler M, Patte-Karsenti N, Thiebaut JB, Gout O, Brandel JP. Tonic spinal cord stimulation as therapeutic option in Parkinson disease with axial symptoms: Effects on walking and quality of life. Parkinsonism Relat Disord. 2019 Jun;63:235-237. doi: 10.1016/j.parkreldis.2019.02.044. Epub 2019 Mar 2. PMID 30852148